CLINICAL TRIAL: NCT04007549
Title: Tobacco and Alcohol Risk Reduction for Women Treated for Breast Cancer and Partner Involvement : Benefits of a Brief Motivational Couple-based Intervention.
Brief Title: Brief Intervention for Tobacco and Alcohol Risk Reduction for Couple During Breast Cancer Treatment.
Acronym: IBMC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal organisation reason
Sponsor: Institut Bergonié (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IB 2017-05; 2017-A03315-48 (Other: Agence nationale de sécurité du médicament et des produits de santé (ANSM))
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Smoking Cessation; Alcohol Use, Unspecified
Keywords: Breast cancer; Smoking cessation; Alcohol risk reduction; Couple intervention; Screening; Brief intervention; Referral to treatment; Randomized Trial
MeSH Terms: conditions — Breast Neoplasms; Smoking Cessation; Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Screening, Brief Intervention and Referral to Treatment (SBIRT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual brief motivational intervention (Experimental): Individual brief motivational intervention (IBMI) on tobacco/alcohol risk reduction for the breast cancer patient; the partner receive e-mail or postal brief advices.
  Interventions: Behavioral: Brief motivational interview on tobacco/alcohol risk reduction
- Couple-based brief motivational intervention (Active Comparator): Couple-based brief motivational intervention (CBMI) on tobacco/alcohol risk reduction.
  Interventions: Behavioral: Brief motivational interview on tobacco/alcohol risk reduction

INTERVENTIONS:
Behavioral: Brief motivational interview on tobacco/alcohol risk reduction — The intervention is a couple brief motivational interview (CBMI) on tobacco/alcohol risk reduction, delivered in a single session and a booster session one month later.
  It is based on motivational interviewing principals (patient-centered communication, expression of empathy, develops discrepancy, deal with resistance to change, support self-efficacy and autonomy), with feedback on tobacco / alcohol consumption, information delivery and if needed referral to treatment. The intervention also specifically focuses on relational dynamics, and marital support development. This intervention will be compared with a single individual brief motivational intervention (IBMI) and a booster session one month later, only delivered to the patient; and the partner receive e-mail or postal brief advices.
  All brief interventions will be carried out by the same psychologist trained and supervised for this type of intervention.

SUMMARY:
This study will examine the benefits of involving partner in a Screening, Brief Intervention and Referral to Treatment (SBIRT) program for tobacco and alcohol for women treated for breast cancer. Using a two-arm randomized trial (couple brief motivational intervention (CBMI) versus individual brief motivational intervention (IBMI) with repeated measures at 6 weeks, 3 and 6 months.

DETAILED DESCRIPTION:
Background: Breast cancer is a common disease for which over 80% of women treated will still be in remission five years after diagnostic. They are a population that can benefit from support to reduce the risks associated with tobacco and alcohol consumptions. Moreover, it is well documented that health behaviors are part of a relational context. Thus, intervene on an individual level cannot suffice to apprehend health behaviors from a systemic perspective. Screening Brief Intervention and Referral to Treatment (SBIRT) program are evaluated for many years and are the reference model in health setting. However, despite national and international recommendations, SBIRT implementation in clinical routine is still very limited in oncology setting. Furthermore, intervene on multiple risk behaviors (contributing to many cancers, increasing the risk of second cancer, treatment morbidity and the risk of developing other chronic diseases) is recommended by several recent empirical studies. Involving the partner in the prevention process could help to develop healthy living environments. A SBIRT program, specifically dedicated to the oncological context and involving the partner may help to reduce tobacco and alcohol risk consumption. Methods/design: The study is a two-arm randomized trial including smoking couples. The intervention is a couple brief motivational intervention (CBMI) on tobacco/alcohol risk reduction, delivered in a single session and a booster session one month later. This intervention will be compared with an individual brief motivational intervention (IBMI) consisting a single brief motivational intervention and a booster session one month later, only delivered to the breast cancer patient; and the partner receive e-mail or postal brief advices. Measures are repeated at 6 weeks, 3 and 6 months post-intervention. The primary outcome is tobacco 7-day point prevalence abstinence (PPA) at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* for the breast cancer patient: patients treated for a first breast cancer; Karnofsky Index> 70;
* for both patient and partner: ≥18 years old; smoking more than or equal to 1 cigarette/day;
* without ongoing treatment for current substance-related disorders; having a good understanding of the French language;
* able to express consent to benefit from intervention focused on smoking cessation;
* having an email address and internet access at home.

Exclusion Criteria:

* Refusal of the patient that his/her partner participates or refusal of the partner to participate
* Individual deprived of liberty, under guardianship or trusteeship
* Individual with a dementia or psychiatric disorder that could compromise informed consent and commitment in different times of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Tobacco 7-day point prevalence abstinence (PPA) at 6 months | 6 months

SECONDARY OUTCOMES:
Tobacco 7-day point prevalence abstinence (PPA) at 6 months | 6 weeks
Tobacco 7-day point prevalence abstinence (PPA) at 6 months | 3 months
Quality of life as per EORTC QLQ-C30 | 6 months
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 - Aaronson et al. JNCI 1993
Quality of life as per EORTC QLQ-C30 | 6 weeks
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 - Aaronson et al. JNCI 1993
Quality of life as per EORTC QLQ-C30 | 3 months
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 - Aaronson et al. JNCI 1993
Nicotine dependence measured using the Fageström (1978) test | 6 months
Nicotine dependence measured using the Fageström (1978) test | 6 weeks
Nicotine dependence measured using the Fageström (1978) test | 3 months
Alcohol consumption based on the AUDIT scale | 6 months
  Alcohol Use Disorders Test short version - Saunders JB, Aasland OG, Babor TF, de la Fuente JR and Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption II. Addiction 1993; 88:791-804.
Alcohol consumption based on the AUDIT scale | 6 weeks
  Alcohol Use Disorders Test short version - Saunders JB, Aasland OG, Babor TF, de la Fuente JR and Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption II. Addiction 1993; 88:791-804.
Alcohol consumption based on the AUDIT scale | 3 months
  Alcohol Use Disorders Test short version - Saunders JB, Aasland OG, Babor TF, de la Fuente JR and Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption II. Addiction 1993; 88:791-804.
Psychological distress Symptom Checklist-90-R | 6 months
  SCL-90-R, Derogatis et al. Psychopharmacol Bull. 1973.
Psychological distress Symptom Checklist-90-R | 6 weeks
  SCL-90-R, Derogatis et al. Psychopharmacol Bull. 1973.
Psychological distress Symptom Checklist-90-R | 3 months
  SCL-90-R, Derogatis et al. Psychopharmacol Bull. 1973.
Scores of conjugal adaptability and cohesion with The Family Adaptability and Cohesion Evaluation Scale (FACE III). | 6 months
Scores of conjugal adaptability and cohesion with The Family Adaptability and Cohesion Evaluation Scale (FACE III). | 6 weeks
Scores of conjugal adaptability and cohesion with The Family Adaptability and Cohesion Evaluation Scale (FACE III). | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Bergonie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No